CLINICAL TRIAL: NCT01286506
Title: Observational Study Evaluating the Hemodynamic Relationship Between Volume Removal and Pulse Pressure Variation During Renal Replacement Therapy
Brief Title: Observational Study of Blood Pressure Measurements and Continuous Dialysis
Status: Terminated | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 16710A; NCT01153087 (obsolete NCT alias)
Record Dates: First submitted 2011-01-27; First posted 2011-01-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Kidney Failure; Respiratory Failure; Critical Illness; Shock
Keywords: Pulse pressure variation; Continuous venovenous hemodialysis; Volume status; Critical care
MeSH Terms: conditions — Renal Insufficiency; Respiratory Insufficiency; Critical Illness; Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Mechanically ventilated patients
- Non-mechanically ventilated patients

SUMMARY:
Dialysis is used to control the fluid balance and metabolic state of patients with kidney disease. Control of the metabolic state, via electrolytes, can be monitored using labs that are routinely drawn from patients undergoing continuous hemodialysis. Control of fluid removal is much more difficult. This study aims to determine whether changes in the blood pressure associated with breathing correlate with or predict intolerance to fluid responsiveness with continuous dialysis.

We hypothesize that a measurement of changes in blood pressure with breathing called arterial pulse pressure variation may be able to predict the ability to remove fluid during continuous renal replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* age > 17 years old
* CVVHD renal replacement therapy
* indwelling arterial line

Exclusion Criteria:

* age < 18 years old
* pregnancy
* temperature < 34°C
* severe mechanical ventilator dyssynchrony
* cardiac arrhythmias precluding automated PPV measurement by ICU monitors
* non-pulsatile cardiac flow
* open thoracic cavity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ICU patients requiring CVVHD who have an indwelling arterial line.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2011-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Predictive value of pulse pressure variation for tolerance of fluid removal on CVVHD | Iterative 24 hr periods for the duration of CRRT

SECONDARY OUTCOMES:
Increased doses of vasoactive agents on CRRT | Iterative 24 hr periods for the duration of CRRT
Inability to meet goal ultrafiltration rate | Iterative 24 hr periods for the duration of CRRT
Hypotensive events on CRRT | Iterative 24 hr periods for the duration of CRRT

CONTACTS AND LOCATIONS:
Overall Officials: Michael O'Connor, MD, Principal Investigator — University of Chicago; Jay L Koyner, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago Medical Center, Chicago, Illinois, United States